CLINICAL TRIAL: NCT02829164
Title: Tonsillectomy and Primitive IgA Nephropathy in Children: Strasbourg Cohort and Assessment Practices in Inter North East Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6402
Record Dates: First submitted 2016-06-16; First posted 2016-07-12 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Tonsillectomy
Keywords: Tonsillectomy; primary IgA nephropathy; primary nephropathy; IgA; Berger's disease; Purpura rheumatoid; kidney failure
MeSH Terms: conditions — Glomerulonephritis, IGA; IgA Vasculitis; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primitive kidney disease IgA, represented by Berger's disease and rheumatoid purpura nephropathy, are the first cause of kidney failure from chronic glomerulonephritis: changes in 20 years to end-stage renal failure is described in 10 to 30 % of cases in Berger's disease and in 15 to 20% of cases in nephropathy HSP. These two pathological entities share biological and histological characteristics, as well as common pathophysiological mechanisms, particularly the production of abnormally glycosylated IgA1 promoting their proliferation in the mesangium. Tonsils part of Iga abnormal production sites that would be associated with an infectious stimulus, tonsillectomy has been studied as a possible treatment in primitive IgA nephropathy. The benefit of tonsillectomy is controversial: many Japanese studies demonstrate its effectiveness in terms of reduction of proteinuria, improved renal function in the long term regression of histological lesions and reduced risk of relapse following clinical remission whereas European studies do not suggest its effectiveness in treating IgA nephropathy. In this context, the aim of our study is to describe the scope of practice of tonsillectomy in the treatment of primary renal disease in IgA child in the inter East region and describe the short renal become Strasbourg end of the cohort that received this treatment.

ELIGIBILITY:
Inclusion criteria:

* Children with a clinical diagnosis and / or histological evidence of primary IgA nephropathy
* Follow the University Hospital of Strasbourg since 2009
* Having received a tonsillectomy in their care
* Children whose holders of parental authority does not oppose the use of clinical data from their child for research purposes

Exclusion criteria:

* Children whose holders of parental authority are opposed to the use of clinical data from their child for research purposes

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with a clinical diagnosis and / or histological evidence of primary IgA nephropathy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the management of the tonsillectomy at the CHU of Strasbourg by a standardized questionnaire | since January 2009

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia HIGEL, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Pédiatrie 1 Hôpital de Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No